CLINICAL TRIAL: NCT06633822
Title: Crown Lengthening in Aesthetic Anterior Sector by Means of Guided Digital Planning: 12-month Randomized Controlled Clinical Trial Comparing the Efficacy of Digital Versus Analog Protocol.
Brief Title: Crown Lengthening in Aesthetic Anterior Sector by Means of Guided Digital Planning: Ramdomized Controlled Clinical Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 24/160-E
Record Dates: First submitted 2024-07-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-02

CONDITIONS: Insufficient Clinical Crown Length
Keywords: Crown lengthening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital plannig (Experimental)
  Interventions: Diagnostic Test: Digital planning
- Analogic planning (Active Comparator)
  Interventions: Diagnostic Test: Analogic planning

INTERVENTIONS:
Diagnostic Test: Digital planning — The digital methodology will consist of obtaining a digital scan and a computed tomography (CBCT) that will be aligned using a digital program for the elaboration of a digital wax-up and fabrication of a printed surgical template.
  Arms: Digital plannig
Diagnostic Test: Analogic planning — The analog wax-up will be elaborated based on a silicone impression and periapical radiographs with parallel technique, which will allow us to elaborate an essix-type surgical splint.
  Arms: Analogic planning

SUMMARY:
The objective of this research is to compare the diagnostic accuracy in the detection of the cementoenamel junction (CEJ) and alveolar bone ridge using guided digital planning versus conventional analog planning for patients with excessive gingival exposure in the smile (gummy smile) due, at least in part, to altered passive eruption.

DETAILED DESCRIPTION:
Forty-four subjects will be randomly assigned to the planning groups according to a digital methodology, DM (n=22) or an analog methodology AM (n=22). Surgical guides will be developed to establish the location of the acementoenamel junction and bone crest. The digital methodology will consist of obtaining a digital scan and a computed tomography (CBCT) that will be aligned using a digital program for the elaboration of a digital wax-up and fabrication of a printed surgical template. The analog wax-up will be elaborated based on a silicone impression and periapical radiographs with parallel technique, which will allow us to elaborate an essix type surgical splint. Measurements will be recorded at baseline, on the day of surgery, at 4, 6 and 12 months of follow-up. Variables related to the patient's experience will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Presence of teeth in the second sextant (edentulous section of a single tooth with the presence of adjacent teeth on both sides of the absence is accepted).
* No sites with attachment loss (AL) > 3 mm in the area to be treated (second sextant).
* Present full mouth plaque index (Ainamo and Bay, 1975) <15%.
* Have bleeding on probing (BoP; Ainamo & Bay 1975) <15%.

Exclusion Criteria:

* pregnancy or lactation
* patients who smoke
* patients under treatment with antimicrobials and anti-inflammatory drugs in the last 2 months or with medications associated with changes in the gingival tissue (antiepileptics, calcium channel blockers, etc.)
* subjects with systemic conditions that alter the normal presentation of the gingival tissue (hereditary gingival fibromatosis) or those diagnosed with uncontrolled diabetes mellitus
* patients with severe dental malposition and/or presence of dental implants in the area to be treated
* use of orthodontic appliances
* all those who present a disability or mental disorders that make it difficult for the patient to understand or follow them during the study period. study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The accuracy of surgical guide. | 12 months
  The accuracy of surgical guide to detect the cementoenamel junction and position of the alveolar bone crest: distance from the splint margin to the CEJ measured intra-surgically in mm at 3 points per tooth using a CP-15 periodontal probe (Hu Friedy®, Leimen, Germany).

SECONDARY OUTCOMES:
The stability of the crown length | 12 months
  The stability of the crown length established over a 12-month period (tissue rebound) measured at 3 points per tooth with a CP-15 millimeter periodontal probe and by intraoral digital scanning.
Patient's phenotype | 12 months
  Therapeutic response according to the patient's phenotype, based on the transparency of the periodontal probe CP-15 (Hu Friedy®, Leimen, Germany) through the gingival margin while probing the buccal sulcus, according to the classification of Rouck et al 2009.
The number of teeth and patients in which the second phase was necessary. | 12 months
  The number of teeth and patients in which the second phase was necessary and the amount of removal of keratinized tissue (gingivectomy) in the second phase (at 4 months) in millimeters using a CP-15 millimeter periodontal probe.
The time spent | 12 months
  The time spent in digital/analog recording in minutes.
Patient satisfaction | 12 months
  Patient satisfaction according to the validated survey (Oral Health Impact Profile OHIP-14).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Dentistry department, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No